CLINICAL TRIAL: NCT00562133
Title: Effect of Prandial Treatment With Insulin Glulisine Compared to Regular Human Insulin on Postprandial Endothelial Function and Microvascular Stress in Type 2 Diabetic Patients
Brief Title: Effect of Insulin Glulisine vs Regular Human Insulin on Postprandial Endothelial Function in Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IKFE Institute for Clinical Research and Development (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: APIDR_L_01896; EudraCT Number 2006-005127-42
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2007-11-21 (Estimated); Status verified 2007-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — insulin glulisine; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): One Day Treatment with Insulin Glulisine
  Interventions: Drug: Insulin Glulisine
- 2 (Active Comparator): One day Treatment with Human insulin
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin Glulisine — 100 IU/ml, 0.10 U/kg immediately before ingestion of a standardised liquid meal
  Other Names: Apidra
  Arms: 1
Drug: Insulin — 100 IU/ml, 0.10 U/kg 15 Minutes before ingestion of a standardised liquid meal
  Other Names: Insuman
  Arms: 2

SUMMARY:
The primary objective of the study is to evaluate the postprandial time course of nitrotyrosine after injection of insulin glulisine compared with regular human insulin.

The secondary objectives are to evaluate the postprandial time course of the following efficacy parameters after injection of insulin glulisine compared with regular insulin on

* Blood Glucose
* Insulin
* Intact proinsulin
* Asymmetric dimethylarginine (ADMA)
* Metal matrix proteasis (MMP-9)
* Oxidative status (per ox)
* Interleukin 18 (IL-18)
* Free fatty acids (FFA)
* Oxidised LDL (ox-LDL)
* Microvascular blood circulation measured with laser Doppler at 37 °C (LDF37)
* Microvascular blood circulation measured with laser Doppler at 44 °C (LDF44)

DETAILED DESCRIPTION:
Phase III b Indication Type 2 Diabetes Trial Objectives 1) Primary objective: The primary objective of the study is to evaluate the postprandial time course of nitrotyrosine after injection of insulin glulisine compared with regular human insulin. 2) Secondary objectives: The secondary objectives are to evaluate the postprandial time course of blood glucose, insulin, intact proinsulin, asymmetric dimethylarginine (ADMA), metal matrix proteasis (MMP-9), free fatty acids (FFA), oxidised LDL (ox-LDL), oxidative status (per ox), IL-18 as well as postprandial time course of microvascular blood circulation measured with laserdopplerflux at 37 °C (LDF37) and 44 C (LDF44).

Efficacy Variables Primary efficacy variablePostprandial time course of nitrotyrosineSecondary efficacy variablePostprandial time course of glucose, insulin, intact proinsulin, ADMA, MMP-9, FFA, ox-LDL, per-ox, and IL-18 as well as postprandial time course of laserdopplerflux at 37 °C and 44 °C Safety Variables Incidence and frequency of adverse events and evaluation of safety laboratory parameters Medication/Dosage Insulin glulisine, dose 0.10 U/kg and Regular Human Insulin, dose 0.10 U/kg Study Duration Duration of study participation for one patient: 5 - 43 days Overall duration of the study: 6 months Design Single-centre, open label, randomized, 2-way-crossover trial Population Male and female type 2 diabetic patients between 40 and 70 years with HbA1c between 6.5 % and 9.9 % and treated with sulfonyurea alone or in combination with Metformin in a stable dosage within the last 3 months Sample Size N = 15

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 Diabetes mellitus according to the ADA criteria
2. HbA1c between 6.5 % and 9.9 %
3. Monotherapy with sulfonylurea or combined with Metformin in a stable dosage within the last 3 months
4. Age between 40 and 70 years
5. BMI < 40

Exclusion Criteria:

1. Type 1 Diabetes mellitus
2. Pre-Treatment with insulin within the last 6 months prior to screening
3. Treatment with glitazones within the last 6 months prior to screening
4. Pre-Treatment with PPARy-agonists, glinides or glucosidase inhibitors within the last 4 weeks prior to screening
5. Untreated hypertension stage II-III according to WHO criteria
6. Planned or anticipated change in antidiabetic and/or concomitant medication during study participation
7. Total Cholesterol > 300 mg/dl (anamnestically)
8. Hypokalemia (K < 3.5 mmol /l)
9. Major micro- or macrovascular complications as judged by the investigator
10. Tobacco use within the last 12 months prior to screening
11. Drugs with major impact on endothelial function like nitrates etc.
12. History of drug or alcohol abuse within the last five years prior to screening
13. Anamnestic history of hypersensitivity to the study drugs or to drugs with similar chemical structures
14. History of severe or multiple allergies
15. Treatment with any other investigational drug within 3 months prior to screening
16. Progressive fatal disease
17. History of significant cardiovascular, respiratory, gastrointestinal, hepatic (ALAT and/or ASAT > 3 times the normal reference range), renal (creatinine > 1.1 mg/dL in women, > 1.5 mg/dL in men), neurological, psychiatric and/or haematological disease as judged by the investigator
18. Pregnancy or breast feeding
19. Sexually active women of childbearing potential not consistently and correctly practicing birth control by implants, injectables, combined oral contraceptives, hormonal intrauterine devices (IUDs), sexual abstinence or vasectomised partner
20. Lack of compliance or other similar reason, that according to investigator, precludes satisfactory participation in the study

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-12; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
the postprandial time course of nitrotyrosine after injection of insulin glulisine compared with regular human insulin | 1 day

SECONDARY OUTCOMES:
postprandial time course of blood glucose, insulin, intact proinsulin, ADMA, MMP-9, FFA, ox-LDL, per ox Status, IL-18, postprandial time course of microvascular blood circulation measured with laserdopplerflux at 37 °C and 44 C | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Forst, Prof, MD, Principal Investigator — Institute for Clinical Research and Development
Locations (1):
- Ikfe, Mainz, Rhineland-Palatinate, Germany